CLINICAL TRIAL: NCT04955249
Title: Impact of Dexmedetomidine Supplemented Analgesia on Delirium and Long-term Outcomes in Elderly After Hip Fracture Surgery: A Multicenter, Double-blinded, Randomized Controlled Trial
Brief Title: Dexmedetomidine Supplemented Analgesia and Delirium After Hip Fracture Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped prematurely because of too few cases.
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-199
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Elderly; Hip Fracture Surgery; Patient-controlled Analgesia; Dexmedetomidine; Postoperative Delirium
Keywords: Elderly; Hip fracture surgery; Patient-controlled analgesia; Dexmedetomidine; Postoperative delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients in this group receive dexmedetomidine-supplemented patient-controlled analgesia for up to 3 days after surgery. The formula is a mixture of dexmedetomidine (1 microgram/ml) and sufentanil (1 microgram/ml), diluted with normal saline to 200 ml. The analgesic pump is programmed to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml at each time and a lockout interval of 8 minutes.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients in this group receive routine patient-controlled analgesia for up to 3 days after surgery. The formula is a mixture of placebo and sufentanil (1 microgram/ml), diluted with normal saline to 200 ml. The analgesic pump is programmed to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml at each time and a lockout interval of 8 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in this group receive dexmedetomidine-supplemented patient-controlled analgesia for up to 3 days after surgery. The formula is a mixture of dexmedetomidine (1 microgram/ml) and sufentanil (1 microgram/ml), diluted with normal saline to 200 ml. The analgesic pump is programmed to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml at each time and a lockout interval of 8 minutes.
  Other Names: Intervention group
  Arms: Dexmedetomidine group
Drug: Placebo — Patients in this group receive routine patient-controlled intravenous analgesia for up to 3 days after surgery. The formula is a mixture of placebo and sufentanil (1 microgram/ml), diluted with normal saline to 200 ml. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml at each time and a lockout interval of 8 minutes.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Delirium is common in the elderly after hip fracture surgery, and is associated with worse outcomes. The investigators hypothesize that, for elderly patients after hip fracture surgery, dexmedetomidine supplemented analgesia can reduce the incidence of delirium and improve the long-term outcomes.

DETAILED DESCRIPTION:
Delirium is a common complication in patients after hip fracture surgery and is associated with worse outcomes, including prolonged hospital stay, poor functional recovery, decreased cognitive function, increased health care costs, and elevated mortality rate.

The etiology of delirium is multifactorial and include severe pain and sleep disturbances after surgery, as well as surgery-related inflammation. Dexmedetomidine is a selective alpha 2 receptor agonist. It exerts sedative effects by activating the endogenous sleep-promoting pathway and leads to a state like non-rapid eye movement sleep. It produces analgesic effects by activating the alpha2a adrenergic receptor subtype in the spinal cord. Perioperative dexmedetomidine also alleviates the degree of surgery-related inflammation.

Previous studies showed that, for elderly patients admitted to the intensive care unit after non-cardiac surgery, low-dose dexmedetomidine infusion improved subjective sleep quality and reduced delirium early after surgery; it also increased survival up to 2 years and improved life quality in 3-year survivors. The investigators hypothesize that dexmedetomidine supplemented patient-controlled analgesia can also reduce delirium and improve long-term outcomes in elderly patients after hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years but < 90 years;
* Scheduled to undergo hip fracture surgery;
* Planned to use patient-controlled intravenous analgesia (PCIA) after surgery.

Exclusion Criteria:

* Refuse to participate in this study;
* Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
* Inability to communicate in the preoperative period because of coma, profound dementia or language barrier;
* Preoperative obstructive sleep apnea (diagnosed sleep apnea syndrome or a STOP-Bang score ≥3 combined with a serum bicarbonate ≥28 mmol/L);
* Sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
* Severe hepatic dysfunction (Child-Pugh class C);
* Severe renal dysfunction (requirement of renal replacement therapy before surgery);
* American Society of Anesthesiologists physical status >IV, or estimated survival ≤24 h.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium within the first 5 days after surgery | Up to 5 days after surgery
  Delirium is assessed twice daily (8:00-10:00 am, 18:00-20:00 pm) with the 3-minute Diagnostic Confusion Assessment Method (3D CAM, for patients without mechanical ventilation) or the Confusion Assessment Method for the intensive care unit (CAM-ICU, for patients with mechanical ventilation) during postoperative days 1-5.

SECONDARY OUTCOMES:
Daily prevalence of delirium during the first 5 days after surgery | Up to 5 days after surgery
  Delirium is assessed twice daily (8:00-10:00 am, 18:00-20:00 pm) with the 3-minute Diagnostic Confusion Assessment Method (3D CAM, for patients without mechanical ventilation) or the Confusion Assessment Method for the intensive care unit (CAM-ICU, for patients with mechanical ventilation) during postoperative days 1-5.
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of non-delirium complications within 30 days after surgery | Up to 30 days after surgery
  Non-delirium complications are defined as new-onset medical events other than delirium that are harmful to patients' recovery and required therapeutic intervention, i.e., grade II or above on the Clavien-Dindo classification.
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality
Quality of life at 30 days | At the 30th day after surgery
  Quality of life is assessed with the WHOQOL-BREF, a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function.
Cognitive function at 30 days | At the 30th day after surgery
  Cognitive function is assessed with the TICS-m, a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 50, with higher score indicating better function.
Overall survival for up to 3 years after surgery | Up to 3 years after surgery
  Time from surgery to all-cause death
Event-free survival for up to 3 years after surgery | Up to 3 years after surgery
  Time from surgery to new-onset diseases or all-cause death, whichever comes first. New-onset disease indicates those that required hospital admission and/or interventional procedures.
Quality of life in 1-，2- and 3-year survivors after surgery | At the end of the 1st, 2nd, and 3rd year after surgery
  Quality of life is assessed with the WHOQOL-BREF, a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function.
Cognitive function in 1-，2- and 3-year survivors after surgery | At the end of the 1st, 2nd, and 3rd year after surgery
  Cognitive function is assessed with the TICS-m, a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 50, with higher score indicating better function.

OTHER OUTCOMES:
Cumulative sufentanil consumption within 5 postoperative days | Up to 5 days after surgery
  Cumulative sufentanil consumption within 5 postoperative days
Pain severity during postoperative days 1-5 | Up to 5 days after surgery
  Pain severity is assessed with twice daily the Numeric Rating Scale (NRS), an 11 point scale where 0=no pain and 10=the worst possible pain.
Subjective sleep quality during postoperative days 1-5 | Up to 5 days after surgery
  Subjective sleep quality is assessed once daily with the Numeric Rating Scale (NRS), an 11 point scale where 0=the best sleep and 10=the worst sleep.
Sedation level during postoperative days 1-5 | Up to 5 days after surgery
  Sedation level is assessed twice daily with the Richmond Agitation-Sedation Scale (RASS), of which the range is as follows: +4 (combative), +3 (very agitated), +2 (agitated), +1 (restless), 0 (alert and clam), -1 (drowsy), -2 (light sedation), -3 (moderate sedation), -4 (deep sedation), and -5 (unarousable).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Zhao X, Dong T, Yang Z, Zhang Q, Zhang Y. Risk factors for postoperative delirium following hip fracture repair in elderly patients: a systematic review and meta-analysis. Aging Clin Exp Res. 2017 Apr;29(2):115-126. doi: 10.1007/s40520-016-0541-6. Epub 2016 Feb 12. PMID 26873816
- [Background] Malik AT, Quatman CE, Phieffer LS, Ly TV, Khan SN. Incidence, risk factors and clinical impact of postoperative delirium following open reduction and internal fixation (ORIF) for hip fractures: an analysis of 7859 patients from the ACS-NSQIP hip fracture procedure targeted database. Eur J Orthop Surg Traumatol. 2019 Feb;29(2):435-446. doi: 10.1007/s00590-018-2308-6. Epub 2018 Sep 18. PMID 30229446
- [Background] Cole MG. Delirium in elderly patients. Am J Geriatr Psychiatry. 2004 Jan-Feb;12(1):7-21. PMID 14729554
- [Background] Mu DL, Zhang DZ, Wang DX, Wang G, Li CJ, Meng ZT, Li YW, Liu C, Li XY. Parecoxib Supplementation to Morphine Analgesia Decreases Incidence of Delirium in Elderly Patients After Hip or Knee Replacement Surgery: A Randomized Controlled Trial. Anesth Analg. 2017 Jun;124(6):1992-2000. doi: 10.1213/ANE.0000000000002095. PMID 28525512
- [Background] Kalisvaart KJ, de Jonghe JF, Bogaards MJ, Vreeswijk R, Egberts TC, Burger BJ, Eikelenboom P, van Gool WA. Haloperidol prophylaxis for elderly hip-surgery patients at risk for delirium: a randomized placebo-controlled study. J Am Geriatr Soc. 2005 Oct;53(10):1658-66. doi: 10.1111/j.1532-5415.2005.53503.x. PMID 16181163
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Weinstein SM, Poultsides L, Baaklini LR, Morwald EE, Cozowicz C, Saleh JN, Arrington MB, Poeran J, Zubizarreta N, Memtsoudis SG. Postoperative delirium in total knee and hip arthroplasty patients: a study of perioperative modifiable risk factors. Br J Anaesth. 2018 May;120(5):999-1008. doi: 10.1016/j.bja.2017.12.046. Epub 2018 Mar 9. PMID 29661417
- [Background] Ravi B, Pincus D, Choi S, Jenkinson R, Wasserstein DN, Redelmeier DA. Association of Duration of Surgery With Postoperative Delirium Among Patients Receiving Hip Fracture Repair. JAMA Netw Open. 2019 Feb 1;2(2):e190111. doi: 10.1001/jamanetworkopen.2019.0111. PMID 30794305